CLINICAL TRIAL: NCT03542422
Title: An Exploratory and Open Clinical Study of Apatinib Mesylate as First-line Treatment for Advanced Esophagus Cancer.
Brief Title: Apatinib as First -Line Treatment for Advanced Esophagus Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-EC-201804
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Advanced Esophagus Cancer
MeSH Terms: interventions — apatinib; tyrosyl-glutamyl-tryptophan; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib (Experimental): Apatinib 500 mg,po,qd,continuous dosing until PD, death or not tolerated toxicity.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Metastasis after primary treatment : Apatinib + yew + platinum. Local recurrence after previous surgery/radiotherapy: Apatinib alone or in combination with platinum-based chemotherapy.
  Other Names: yew; platinum

SUMMARY:
An Exploratory study of Amapinib for patients with advanced esophagus cancer .

DETAILED DESCRIPTION:
An Exploratory study of Amapinib for patients with advanced esophagus cancer .

Eligible are patients with advanced esophagus cancer. Apatinib (500mg) is given daily as follows:

Metastasis after primary treatment : Apatinib + yew + platinum. Local recurrence after previous surgery/radiotherapy: Apatinib alone or in combination with platinum-based chemotherapy One therapy cycle has 28 days. Tumor response is evaluated every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 to 75 years old, men and women;
* 2. Patients diagnosed with esophageal squamous cell carcinoma by histopathology and immunohistochemistry;
* 3. ECOG performance status: 0-2;
* 4. Life expectancy ≥ 12 weeks;
* 5. Clinical stage IIIb-IV; metastatic patients who have not initially received chemotherapy or patients who have local recurrence after surgery or radiochemotherapy (no local treatment indication) ;
* 6. Function of the major organs is normal, criteria referred are as follow:

  1. blood routine examination: HB ≥ 90g/L (no blood transfusion within 14 days); ANC ≥ 1.5 × 109/L; PLT ≥ 80 × 109/L;
  2. biochemical examination: ALB ≥ 29 g / L (AlB did not lose within 14 days); ALT and AST <5 ULN; TBIL ≤ 1.5 ULN;
  3. plasma examination Cr ≤ 1.5 ULN;
* 7. Subjects voluntarily participated in the study, signed informed consent, have good compliance and cooperate with follow-up;
* 8. Patients that the investigator believes can benefit.

Exclusion Criteria:

* 1. Those who have had other malignant tumors in the past or at the same time;
* 2. Pregnant or lactating women;
* 3. Patients with high blood pressure and can't get a good control after antihypertensive drug therapy (systolic blood pressure>150mmHg, diastolic blood pressure>100mmHg); patients with grade Ⅱ or more myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTC interval≥450ms) and Ⅲ~Ⅳ grade cardiac insufficiency according to NYHA; cardiac color Doppler ultrasonography: LVEF <50%;
* 4. Unable to swallow, chronic diarrhea, and intestinal obstruction, which significantly affects drug taking and absorption;
* 5. Have a clear risk of gastrointestinal bleeding concerns (such as local active ulcer lesions, fecal occult blood + or more), a history of gastrointestinal bleeding within 6 months;
* 6.With coagulation abnormalities (PT>16 s, APTT>43 s, TT>21 s, Fbg <2 g/L), hemorrhagic tendency or receiving thrombolysis or anticoagulant therapy;
* 7. Have a mental illness, or history of abuse of psychotropic substances;
* 8. With anastomotic recurrence and tracheal fistula;
* 9. Patients who participated in other drug clinical trials within 4 weeks;
* 10. Patients who have concomitant diseases that are seriously compromise the patient's safety or affect the patient to complete the study according to the researcher's judgment;
* 11. Researchers believe that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-30 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Progress free survival（PFS） | 12months
  Time subject into the group to tumor objective progression.

SECONDARY OUTCOMES:
Overall Survival | up to12months
  Time subject into the group to die

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan, China